CLINICAL TRIAL: NCT03075527
Title: A Phase 2 Study of Durvalumab in Combination With Tremelimumab in Malignant Pleural Mesothelioma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Criteria not met for second stage at time of interim analysis
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Biagio Ricciuti, Sponsor Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-549
Record Dates: First submitted 2017-03-02; First posted 2017-03-09 (Actual); Results first posted 2019-11-12 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Mesothelioma
Keywords: Mesothelioma
MeSH Terms: conditions — Mesothelioma | interventions — tremelimumab; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tremelimumab + Durvalumab (Experimental): Subjects will receive durvalumab and tremelimumab both via intravenous infusion once per day for every 28 day cycles (+ 7 days). Participants will receive tremelimumab for up to 4 cycles (4 doses). Beginning with cycle 5 day 1, subjects will continue to receive durvalumab alone, until clinical or radiological progression.
  Interventions: Drug: Tremelimumab; Drug: Durvalumab

INTERVENTIONS:
Drug: Tremelimumab — Tremelimumab blocks a receptor on immune cells that normally suppresses immune attack.
  Other Names: CP-675,206
Drug: Durvalumab — Durvalumab is a drug that blocks a protein often produced by cancer cells or surrounding cells to suppress immune cells from attacking cancer cells.
  Other Names: MEDI-4736

SUMMARY:
This research study is studying a pair of immunotherapies as a possible treatment for malignant pleural mesothelioma.

The drugs involved in this study are:

* Durvalumab
* Tremelimumab

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved durvalumab or tremelimumab as a treatment for any disease.

In this research study, the investigators are studying if the study drug can help your cancer compared to the usual approach to treating malignant pleural mesothelioma . Durvalumab is a drug that blocks a protein often produced by cancer cells or surrounding cells to suppress immune cells from attacking cancer cells. Tremelimumab blocks a receptor on immune cells that normally suppresses immune attack. These two study drugs have been used alone for mesothelioma but the combination has not yet been tested for mesothelioma. These two drugs have been used for cancers such as melanoma and have been effective than using either drug alone.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained prior to any study-specific procedures not considered part of routine medical care
* Histologically or cytologically confirmed unresectable or medically inoperable malignant pleural mesothelioma
* Disease progression after treatment with at least one line of chemotherapy that included a first-line platinum agent in combination with an anti-folate
* Participants must have measurable disease according to modified RECIST for pleural malignant mesothelioma. (Bone metastases are not considered measurable.) Prior radiation to the only site of measurable disease will make the participant ineligible unless the lesion has been demonstrated to grow after completion of radiation therapy.
* Participants must be willing and able to undergo a biopsy at the start of this study and an on-treatment biopsy if safe and feasible.
* Participants must have be at least 28 days from any major surgery.
* ECOG performance status of 0 or 1.
* Subjects must have adequate hematologic, renal, and organ and marrow function
* Age 18 years or older
* Female subjects of childbearing potential who are sexually active with a non sterilized male partner must agree to use at least one highly effective method of contraception from the time of screening and must agree to continue using such precautions for 180 days after the last dose of investigational product. Male partners of a female subject must also agree to use male condom plus spermicide throughout this period. Cessation of birth control after this point should be discussed with a responsible physician. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however, occasional abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception. Female patients should refrain from breastfeeding throughout this period.
* Females of childbearing potential are defined as those who are not surgically sterile (i.e., bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or post-menopausal (defined as greater than or equal to 12 months with no menses without an alternative medical cause)
* Non-sterilized male subjects who are sexually active with a female partner of childbearing potential must use male condom plus spermicide from screening through 180 days after the last dose of investigational product. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however, occasional abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception. Male patients should refrain from sperm donation throughout this period. Female partners of a male subject must use a highly effective method of contraception throughout this period.
* Ability to understand and the willingness to sign a written informed consent document
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up

Exclusion Criteria:

* Previous treatment with an immune check-point inhibitors, CTLA-4, PD-1, or PD-L1, including prior treatment with either durvalumab or tremelimumab
* Known central nervous system metastasis. Patients with known brain metastases, spinal cord compression, carcinomatous meningitis, or leptomeningeal disease may be enrolled if they have been treated, are no longer taking corticosteroids, and have been stable on imaging for at least 3 weeks
* Subjects currently receiving systemic corticosteroids above 10 mg per day for more than 14 days; subjects receiving other systemic immunosuppressive drugs for more than 14 days. Exceptions include: inhaled, intranasal, ophthalmic, and topical corticosteroids, local corticosteroid injections (e.g., intra-articular injections), and subjects requiring corticosteroid pre-medication for hypersensitivity reactions (e.g. CT scan premedication)
* Subjects with medical conditions that require the chronic use of systemic corticosteroids. Exceptions include: inhaled, intranasal, ophthalmic, and topical corticosteroids, local corticosteroid injections (e.g., intra-articular injections), and subjects requiring corticosteroid pre-medication for hypersensitivity reactions (e.g. CT scan premedication)
* Active or prior documented autoimmune disease within the past 2 years, including but not limited to systemic lupus erythematosus, sarcoidosis syndrome, or Wegener's granulomatosis. NOTE: Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment within the past 2 years are not excluded.
* Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis, celiac disease, diverticulitis), or any other chronic, serious gastrointestinal condition associated with diarrhea. NOTE: Subjects with known diverticulosis are permitted to enroll.
* History of interstitial lung disease or pneumonitis that has required steroid administration.
* History of primary immunodeficiency
* History of allogeneic organ transplant
* History of hypersensitivity to tremelimumab, durvalumab, or any excipient
* Known history of active tuberculosis
* Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving durvalumab or tremelimumab
* Participants with a history of a second primary malignancy. Exceptions include: patients with a history of malignancies that were treated curatively and have not recurred within 5 years prior to study entry; resected basal and squamous cell carcinomas of the skin, and completely resected carcinoma in situ of any type.
* Participants who have had chemotherapy, biologic therapy, or investigational therapy within 21 days (including bevacizumab) or radiotherapy within 7 days prior to entering the study or those who have not recovered from adverse events due to agents administered
* Any history of a prior immune-related adverse event (irAE) at least or greater than grade 3 while receiving any previous immunotherapy agent.
* Participants who are receiving any other investigational agents.
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection
  * Gastritis
  * Symptomatic congestive heart failure
  * Severe hypertension (defined as BP at least or greater than160/100 during the screening period despite optimal medical management)
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Active bleeding diatheses
  * Active peptic ulcer disease
  * Psychiatric illness/social situations that would limit compliance with study requirements
* Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Fredericia's Correction
* Known past or present medical history HIV-positive
* Subjects with known acute or chronic hepatitis B or hepatitis C.
* Pregnant women are excluded from this study because tremelimumab and durvalumab have unknown effects on the developing fetus. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with tremelimumab or durvalumab, breastfeeding women are also excluded. Female subjects of child bearing potential must have a negative serum pregnancy test obtained prior to trial registration.
* Subjects who are involved in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
* Subjects who have undergone a pneumonectomy due to known potential for pulmonary toxicities and heightened risk for complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2019-06-07 (Actual); Study Completion 2024-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark M. Awad, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute; Biagio Ricciuti, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled from April 2017 to August 2018.
Period: Overall Study
Arm/Group | Tremelimumab + Durvalumab
Started | 19
Completed | 0
Not Completed | 19
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 3
Not completed — Progression/Relapse | 14

BASELINE CHARACTERISTICS:
Arm/Group | Tremelimumab + Durvalumab
Number analyzed (Participants) | 19
Age, Customized [Median (Full Range); unit: years]
  Age | 69 [33 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Overall Response Rate (ORR) was defined as the proportion of participants achieving complete response (CR) or partial response (PR) as best response on treatment based on RECIST v1.1 criteria.
Time Frame: ORR was assessed every 8 weeks from Cycle 1 Day 1 until date of documented disease progression or death. The median treatment duration is 1.91 months with range (0.00 months - 23.46 months).
Population: The analysis population is comprised of eligible and treated patients.
Measure: Number (80% Confidence Interval); unit: proportion of paticipants
Arm/Group | Tremelimumab + Durvalumab
Number analyzed (Participants) | 19
proportion of paticipants | 0.105 [0.045 to 0.229]

2. Secondary Outcome: Median Overall Survival (OS)
Description: OS based on the Kaplan-Meier method is defined as the time from study entry to death or censored at date last known alive.
Time Frame: OS is assessed from date of registration until date of death on-treatment or during follow-up. Survival data collection in long-term follow-up every 3-4 months. Median follow-up for survival is of 27.33 months with range (0.76 months - 50.40 months).
Population: The analysis population is comprised of eligible and treated patients.
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Tremelimumab + Durvalumab
Number analyzed (Participants) | 19
months | 9.76 [7.2 to 29.2]

3. Secondary Outcome: Median Progression Free Survival (PFS)
Description: PFS based on the Kaplan-Meier method is defined as the duration between randomization and documented disease progression (PD) defined per RECIST 1.1 criteria. or death, or is censored at time of last disease assessment.
Time Frame: Participants were evaluated for response every 8 weeks on study and in long-term survival followed-up every 3-4 months. Median follow-up for survival is of 27.33 months with range (0.76 months - 50.40 months).
Population: The analysis population is comprised of eligible and treated patients.
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Tremelimumab + Durvalumab
Number analyzed (Participants) | 19
months | 3.42 [2.79 to 5.72]

4. Secondary Outcome: Median Duration of Response (DOR)
Description: DOR is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (or censored at the date of last disease evaluation).
Time Frame: The median of treatment duration is 1.91 months with range (0.00 months - 23.46 months).
Population: This analysis dataset is comprised of all patients who had a CR or PR on treatment.
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Tremelimumab + Durvalumab
Number analyzed (Participants) | 2
months | 2.07 [2.07 to NA] — The upper bound of the 80% CI for median DOR is NA due to insufficient events.

5. Secondary Outcome: Grade 4-5 Treatment-related Toxicity Rate
Description: All grade 4-5 adverse events (AE) with treatment attribution of possibly, probably or definite based on CTCAEv4.03 that are not resolved in accordance with treatment guidelines were counted. Rate is the proportion of treated participants experiencing at least one of these adverse events as defined during the time of observation.
Time Frame: Toxicity is assessed from the time of first dose of study medication until the participant comes off study. The median of treatment duration is 1.91 months with range (0.00 months - 23.46 months).
Population: This analysis dataset is comprised of all eligible and treated patients.
Measure: Number (80% Confidence Interval); unit: proportion of paticipants
Arm/Group | Tremelimumab + Durvalumab
Number analyzed (Participants) | 19
proportion of paticipants | 0.158 [0.061 to 0.322]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of first dose through end of follow-up, every 3 weeks during active therapy. The median of the observation period for all-cause mortality is 27.33 months with range (0.76 months - 50.40 months). The median of observation time for AE is 1.91 months with range (0.00 months - 23.46 months).
Description: A serious adverse event (SAE) is any AE that: results in death, is immediately life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect in offspring of the subject, is an important medical event that may jeopardize the subject or may require medical intervention to prevent one of the outcomes listed above.
Arm/Group | Tremelimumab + Durvalumab
All-Cause Mortality (participants affected / at risk) | 11/19
Serious Adverse Events (participants affected / at risk) | 4/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tremelimumab + Durvalumab (N=19)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Spinal Cord Compression (Musculoskeletal and connective tissue disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Death NOS (General disorders) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tremelimumab + Durvalumab (N=19)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Congenital, familial and genetic disorders - Other, specify (Congenital, familial and genetic disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 3 (3)
Hypothyroidism (Endocrine disorders) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (3)
Chills (General disorders) | 1 (1)
Edema limbs (General disorders) | 3 (3)
Fatigue (General disorders) | 7 (7)
General disorders and administration site conditions - Other, specify (General disorders) | 2 (2)
Localized edema (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2)
Pain (General disorders) | 3 (3)
Lung infection (Infections and infestations) | 1 (1)
Rash pustular (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 2 (2)
Creatinine increased (Investigations) | 3 (3)
Investigations - Other, specify (Investigations) | 2 (2)
Lipase increased (Investigations) | 4 (4)
Neutrophil count decreased (Investigations) | 1 (1)
Serum amylase increased (Investigations) | 3 (3)
Weight gain (Investigations) | 1 (1)
Weight loss (Investigations) | 2 (2)
White blood cell decreased (Investigations) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (3)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 (6)
Hyponatremia (Metabolism and nutrition disorders) | 4 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-12): https://cdn.clinicaltrials.gov/large-docs/27/NCT03075527/Prot_SAP_000.pdf